CLINICAL TRIAL: NCT03451071
Title: Postpartum HPV Vaccination: Acceptability, Uptake and Immunogenicity
Brief Title: Postpartum HPV Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Haller Smith, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 000518236
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: HPV-Related Malignancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gardasil9 (Experimental)
  Interventions: Drug: Gardasil9

INTERVENTIONS:
Drug: Gardasil9 — Gardasil 9

SUMMARY:
Human papillomavirus (HPV)-related cancers are on the rise in the United States. Furthermore, greater than 90% of cervical cancer cases are attributable to HPV, and cervical cancer disproportionately affects women of color in both incidence and mortality. Due to low HPV vaccine uptake in the US, innovative approaches to vaccinating vulnerable populations are necessary in order to maximize the cancer prevention potential of this vaccine. The puerperium is a time period when women are engaged in the healthcare system and have almost universal access to affordable health care. Two prior studies have shown that postpartum HPV vaccination is acceptable to patients, and high rates of vaccination were achieved in these primarily Hispanic populations. However, data show that the immune response in young women is less robust than in adolescents, and no studies have examined immunogenicity in postpartum women specifically. We propose an HPV vaccination pilot study in women who receive postpartum care at University of Alabama at Birmingham (UAB) hospital. We will examine the acceptability, uptake and immunogenicity of the vaccine in the postpartum setting.

ELIGIBILITY:
Inclusion Criteria:

* postpartum day 0-4 after vaginal or Cesarean delivery at UAB hospital

Exclusion criteria

* Fetal demise or miscarriage, autoimmune disorder, HIV, Hepatitis B/C, chronic steroid use, preeclampsia, non-English speaking

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 195 women consented to participate in the study. 139 consented to survey only, 56 consented to survey and Gardasil9 vaccine.
Period: First Vaccine
Arm/Group | Gardasil9
Started | 56
Completed | 55
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Vaccine
Arm/Group | Gardasil9
Started | 55
Completed | 36
Not Completed | 19
Not completed — Lost to Follow-up | 19
Period: Third Vaccine
Arm/Group | Gardasil9
Started | 36
Completed | 14
Not Completed | 22
Not completed — Lost to Follow-up | 22
Period: Final Questionnaire and Blood Draw
Arm/Group | Gardasil9
Started | 14
Completed | 10
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Gardasil9
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (2.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female only | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black | 48
  Hispanic/Latino | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Indication of Willingness to Accept the Vaccine Based on Survey
Description: This was established using a survey to indicate willingness to receive vaccine.
Time Frame: 1 day (at the time of initial recruitment /survey)
Population: 56 patients consented to vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 195
Participants | 56

2. Secondary Outcome: Uptake of the Vaccine Doses
Description: Those that actually received the vaccine and each time point.
Time Frame: at baseline
Population: 1 participant consented to vaccine and then subsequently withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 56
Participants | 55

3. Secondary Outcome: Uptake of the Vaccine Doses
Description: Those that actually received the vaccine and each time point.
Time Frame: at 3 months
Population: 1 patient consented to vaccine and then withdrew
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 55
Participants | 36

4. Secondary Outcome: Uptake of the Vaccine Doses
Description: Those that actually received the vaccine and each time point.
Time Frame: at 6 months
Population: 36 patients received the 2nd vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Gardasil9
Number analyzed (Participants) | 36
Participants | 14

5. Secondary Outcome: Serum Titers of Vaccine-specific HPV Types
Description: Immunogenicity
Time Frame: baseline and 7 months
Population: This data was not collected
Arm/Group | Gardasil9
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Gardasil9
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 1/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil9 (N=55)
Flu-like symptoms (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT03451071/Prot_SAP_000.pdf